CLINICAL TRIAL: NCT04369781
Title: Oximetrie Transcutanee et Ischemie Critique
Brief Title: Critical Limb Ischemia and Transcutaneous Oximetry
Acronym: CITRA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2019-44
Record Dates: First submitted 2020-04-28; First posted 2020-04-30 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-06

CONDITIONS: Critical Limb Ischemia
Keywords: transcutaneous oxygen pressure
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Suspected critical limb ischemia: Patients referred for transcutaneous oxygen pressure measurements due to a clinical suspicion of critical limb ischemia
  Interventions: Diagnostic Test: transcutaneous oxygen pressure recording at rest

INTERVENTIONS:
Diagnostic Test: transcutaneous oxygen pressure recording at rest — Recording of limb and chest transcutaneous oxygen pressure

SUMMARY:
Retrospective analysis of transcutanesou oximetry (Tcpo2) recording for patients referred with suspected critical limb ischemia searching for specific changes in TcpO2 patterns.

DETAILED DESCRIPTION:
* Patients had Tcpo2 recording at the suspected limb and chest level at rest in the lying position.
* Provocative tests (leg elevation, leg lowering, oxygen inhalation) were performed to improve the sensitivity of tests.
* TcpO2 results were recorded on a 1 Hz bais for of line analysis after anonymization.
* We recorded age , gender, weight, height, ongoing treatments , History of cardiac or respiratory disease.

Visual and mathematical analysis of the TcpO2 recording at the chest and limb level searching for various indices of TcpO2 variability at rest, or differences in responses between the chest and limb tcpO2 responses to provocative tests..

ELIGIBILITY:
Inclusion Criteria:

* Referral for suspected critical limb ischemia

Exclusion Criteria:

* Absence of recording, deny to use medical file

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients referred for critical limb ischemia
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-10-15 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Variability of TcpO2 | 1 hour
  Study of TcpO2 variability

CONTACTS AND LOCATIONS:
Overall Officials: Pierre ABRAHAM, MD; PhD, Principal Investigator — University and univerity hospital in Angers, FRANCE
Locations (1):
- University Hospital, Angers, France

IPD SHARING:
Plan to Share IPD: Undecided
Data available under reasonable request to the investigator